CLINICAL TRIAL: NCT04899245
Title: ReSET Aim 1b: Restarting Safe Education and Testing for Children With Medical Complexity - SARS-CoV-2 Testing in School With Children and Staff
Brief Title: ReSET Aim 1b: Restarting Safe Education and Testing for Children With Medical Complexity - COVID-19 Testing in School With Children and Staff
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2021-0488; A536771 (Other: UW Madison); SMPH/PEDIATRICS (Other: UW Madison); Protocol Version 7/11/22 (Other: UW Madison); 1OT2HD107558-01 (NIH); 2022-0810 (Other: UW Madison)
Record Dates: First submitted 2021-05-19; First posted 2021-05-24 (Actual); Results first posted 2024-07-17 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-06

CONDITIONS: Children With Medical Complexity (CMC); COVID-19
Keywords: In-school COVID testing; Caregiver; School staff; In-person school attendance
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: This is a single site study taking place over 24 months and involving (65) caregivers and their children, and (50) school staff.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- School Staff (Experimental): 50 school staff from Waisman Early Childhood Program (WECP) will be recruited to participate in this study. School staff will send a letter to all WECP staff inviting them to participate. Staff new to the school or who initially decline participation and then reconsider may join at any time.
  Additionally, staff who are vaccinated will be asked to participate in testing.
  Interventions: Diagnostic Test: BinaxNOW Rapid Antigen System
- Parent/Child with Children with medical complexity (CMC) (Experimental): 65 children and their parents will be recruited to participate. School staff will send a letter to all parents with children enrolled in the Waisman Early Childhood Program (WECP) inviting them to participate. Families new to the school or who initially decline participation and then reconsider may join at any time. Participants will also be offered the option of as needed symptomatic home testing.
  Additionally, parents who are vaccinated will be asked to participate in testing. Siblings may be enrolled in the study.
  Interventions: Diagnostic Test: BinaxNOW Rapid Antigen System

INTERVENTIONS:
Diagnostic Test: BinaxNOW Rapid Antigen System — BinaxNOW Rapid Antigen System (Abbott) is a point-of-care, lateral flow immunoassay intended for the qualitative detection of nucleocapsid protein antigen from SARS-CoV-2 in direct anterior nasal (nares) swabs. Internal controls are built into the testing system and results are available in 15 minutes.
  The use of the BinaxNOW system is authorized under the Food and Drug Administration's Emergency Use Authorization. The test is allowed for over-the-counter, non-prescription use with or without symptoms. The test may be used with children two years and older with the help of sample collection by an adult, and the test may be self-administered by anyone aged 15 years or more.

SUMMARY:
The Coronavirus Disease 2019 (COVID-19), caused by the SARS-CoV-2 virus, is a worldwide pandemic that has resulted in large-scale quarantines in cities, states, and countries throughout the world. SARS-CoV-2 is a respiratory virus that is most commonly spread via contact with infective respiratory droplets and aerosols produced by coughing, sneezing, talking, and singing.

Children with medical complexity (CMC), i.e., children with multiple severe chronic conditions, high resource use, severe functional limitations, and substantial family-identified service needs, are a medically vulnerable population for the development of severe COVID-19. Deciding to send CMC to school poses a major dilemma to families wanting to minimize severe COVID-19 risk. School personnel also face risks when CMC attend school. Despite these challenges, achieving in-person school attendance is critical for CMC. Compared to non-CMC, academic and social development for most CMC hinges on being at school. Severe intellectual and developmental disability impairs one's ability to engage with online platforms. Health-promoting services delivered at school, e.g., physical, occupational, and speech therapy, are likely less effective when delivered virtually. Parents of CMC, already disproportionately unemployed due to their child's care needs, experience added employment strain when their child is out of school.

The study objective is to increase the safe return to school for CMC by 1) evaluating the feasibility of school-based COVID-19 testing strategies and 2) identifying parent and staff perceptions of testing and school attendance. A related study (ReSET Aim 1a, NCT04895085) will evaluate the same factors in home-based testing strategies in CMC exclusively.

ELIGIBILITY:
Inclusion Criteria:

* Parents and staff must be at least 18 years of age.
* Staff must have a classroom role (e.g., teacher, aide, playground assistant)
* Parents and staff must be proficient in English.
* Parents and staff must have access to a web-enabled device (phone, tablet, or computer).
* Staff, parent and child must be residents of Wisconsin.
* Parent/child must be enrolled at WECP for the 2021 and/or 2022 school year.

Exclusion Criteria:

* Failure to meet all inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2021-05-04 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Coller, MD, MPH, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin School of Medicine and Public Health, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The protocol enrollment, started, and completed values reflect caregiver/child dyads. There were n = 41 caregivers, n = 47 children.
Groups:
- Parent/Caregiver of Children With Medical Complexity (CMC); Child With Medical Complexity: 65 children and their parents will be recruited to participate. School staff will send a letter to all parents with children enrolled in the Waisman Early Childhood Program (WECP) inviting them to participate. Families new to the school or who initially decline participation and then reconsider may join at any time. Participants will also be offered the option of as needed symptomatic home testing.
  Additionally, parents who are vaccinated will be asked to participate in testing. Siblings may be enrolled in the study.
  BinaxNOW Rapid Antigen System: BinaxNOW Rapid Antigen System (Abbott) is a point-of-care, lateral flow immunoassay intended for the qualitative detection of nucleocapsid protein antigen from SARS-CoV-2 in direct anterior nasal (nares) swabs. Internal controls are built into the testing system and results are available in 15 minutes.
  The use of the BinaxNOW system is authorized under the Food and Drug Administration's Emergency Use Authorization. The test is allowed for over-the-counter, non-prescription use with or without symptoms. The test may be used with children two years and older with the help of sample collection by an adult, and the test may be self-administered by anyone aged 15 years or more.
- School Staff: 50 school staff from Waisman Early Childhood Program (WECP) will be recruited to participate in this study. School staff will send a letter to all WECP staff inviting them to participate. Staff new to the school or who initially decline participation and then reconsider may join at any time.
  Additionally, staff who are vaccinated will be asked to participate in testing.
  BinaxNOW Rapid Antigen System: BinaxNOW Rapid Antigen System (Abbott) is a point-of-care, lateral flow immunoassay intended for the qualitative detection of nucleocapsid protein antigen from SARS-CoV-2 in direct anterior nasal (nares) swabs. Internal controls are built into the testing system and results are available in 15 minutes.
  The use of the BinaxNOW system is authorized under the Food and Drug Administration's Emergency Use Authorization. The test is allowed for over-the-counter, non-prescription use with or without symptoms. The test may be used with children two years and older with the help of sample collection by an adult, and the test may be self-administered by anyone aged 15 years or more.
Period: Overall Study
Arm/Group | Parent/Caregiver of Children With Medical Complexity (CMC) | Child With Medical Complexity | School Staff
Started | 41 | 47 (Children were enrolled as caregiver/child dyads where caregiver n = 41 and child n = 47. Several caregivers enrolled multiple children.) | 24
Completed | 17 | 19 (Children were enrolled as caregiver/child dyads where caregiver n = 17 and child n = 19. Several caregivers enrolled multiple children.) | 21
Not Completed | 24 | 28 | 3
Not completed — Withdrawal by Subject | 3 | 5 | 2
Not completed — No longer eligible - Left staff position | 0 | 0 | 1
Not completed — No longer eligible - Child graduated from school program | 19 | 21 | 0
Not completed — No longer eligible - Moved away from area | 2 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Children With Medical Complexity (CMC); Parent/Caregiver With Children With Medical Complexity (CMC): 65 children and their parents will be recruited to participate. School staff will send a letter to all parents with children enrolled in the Waisman Early Childhood Program (WECP) inviting them to participate. Families new to the school or who initially decline participation and then reconsider may join at any time. Participants will also be offered the option of as needed symptomatic home testing.
  Additionally, parents who are vaccinated will be asked to participate in testing. Siblings may be enrolled in the study.
  BinaxNOW Rapid Antigen System: BinaxNOW Rapid Antigen System (Abbott) is a point-of-care, lateral flow immunoassay intended for the qualitative detection of nucleocapsid protein antigen from SARS-CoV-2 in direct anterior nasal (nares) swabs. Internal controls are built into the testing system and results are available in 15 minutes.
  The use of the BinaxNOW system is authorized under the Food and Drug Administration's Emergency Use Authorization. The test is allowed for over-the-counter, non-prescription use with or without symptoms. The test may be used with children two years and older with the help of sample collection by an adult, and the test may be self-administered by anyone aged 15 years or more.
- Total: Total of all reporting groups
Arm/Group | School Staff | Children With Medical Complexity (CMC) | Parent/Caregiver With Children With Medical Complexity (CMC) | Total
Number analyzed (Participants) | 24 | 47 | 41 | 112
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 40 [28 to 47] | 3 [2 to 4] | 36 [34 to 39] | NA [NA to NA] — Child, parent, and staff ages were analyzed separately.
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex: Female | 23 | 20 | 31 | 74
  Sex: Male | 1 | 22 | 9 | 32
  Sex: Not reported | 0 | 5 | 1 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 4 | 1 | 5
  Not Hispanic or Latino | 24 | 39 | 39 | 102
  Unknown or Not Reported | 0 | 4 | 1 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1 | 2
  Asian | 4 | 2 | 3 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 2 | 4
  White | 20 | 32 | 32 | 84
  More than one race | 0 | 5 | 1 | 6
  Unknown or Not Reported | 0 | 5 | 2 | 7
Region of Enrollment [Number; unit: participants]
  United States | 24 | 47 | 41 | 112

OUTCOME MEASURES:

1. Primary Outcome: Change in Protocol Uptake: Number of Children and Staff Consented Compared to Number of Approached
Description: Feasibility of school based COVID-19 testing will be evaluated by protocol uptake. Data will be retrieved from the study log. Two data limitations to note:
  * The enrollment rate was not stratified by caregiver and child number at the time of data collection. The data was collected at the level of the child.
  * The enrollment rate was not stratified by caregiver/child dyad and staff at the time of data collection. This is a limitation of our data. It is not possible to stratify this outcome and it is therefore analyzed together.
Time Frame: Study duration (up to 21 months)
Population: The number analyzed must include those who were approached and not consented in addition to those consented.
Measure: Number; unit: Participants
Groups:
- Staff and Children: The enrollment rate was not stratified by staff and caregiver/child dyad during data collection.
Arm/Group | Staff and Children
Number analyzed (Participants) | 88
Participants
  Number approached, enrolled | 71
  Number approached, not enrolled | 17

2. Primary Outcome: Change in COVID Test Rate at School: Number of Total Child and Staff Tests Completed as Compared to Number of Tests Expected
Description: * Tests expected: Children and staff in this study will have nasal swab testing performed at school twice weekly (as well as anytime they have symptoms) for the first 3 months of the study. After 3 months, the twice-weekly testing may decrease to symptom-only testing if the rate of COVID spread decreases in Wisconsin. Symptom-only testing is not included as an "expected" test.
  * The number of tests expected was assessed specifically for this outcome measure to determine if testing was proceeding as expected. This value was based on the number of children and staff enrolled at a given time, whether surveillance or symptom-only testing was being conducted, and if any of the participants had COVID-19 (excluding them from testing). This value was not created at baseline, but was dynamic over the course of the study dependent upon the aforementioned factors.
  * The tests expected value was not stratified by child and staff at the time of data collection. It is a limitation of the data.
Time Frame: Every week up to 21 months
Measure: Number; unit: BinaxNow Rapid Antigen COVID-19 Tests
Units Other Than Participants: BinaxNOW Rapid Antigen COVID-19 Tests
Groups:
- Children With Medical Complexity (CMC) AND School Staff: Data was not stratified by school staff and child during data collection.
Arm/Group | Children With Medical Complexity (CMC) AND School Staff
Number analyzed (Participants) | 71
Number analyzed (BinaxNOW Rapid Antigen COVID-19 Tests) | 2368
BinaxNow Rapid Antigen COVID-19 Tests
  Number of tests completed | 2368
  Number of tests expected | 2688

3. Primary Outcome: Change in Symptomatic Test Rate: Number of Symptomatic Tests Completed
Description: Data will be retrieved from study log.
Time Frame: Study duration (up to 21 months)
Measure: Number; unit: Symptomatic BinaxNow Rapid Antigen Tests
Units Other Than Participants: BinaxNOW Rapid Antigen COVID-19 Tests
Groups:
- Parent/Child With Children With Medical Complexity (CMC): 65 children and their parents will be recruited to participate. School staff will send a letter to all parents with children enrolled in the Waisman Early Childhood Program (WECP) inviting them to participate. Families new to the school or who initially decline participation and then reconsider may join at any time. Participants will also be offered the option of as needed symptomatic home testing.
  Additionally, parents who are vaccinated will be asked to participate in testing. Siblings may be enrolled in the study.
  BinaxNOW Rapid Antigen System: BinaxNOW Rapid Antigen System (Abbott) is a point-of-care, lateral flow immunoassay intended for the qualitative detection of nucleocapsid protein antigen from SARS-CoV-2 in direct anterior nasal (nares) swabs. Internal controls are built into the testing system and results are available in 15 minutes.
  The use of the BinaxNOW system is authorized under the Food and Drug Administration's Emergency Use Authorization. The test is allowed for over-the-counter, non-prescription use with or without symptoms. The test may be used with children two years and older with the help of sample collection by an adult, and the test may be self-administered by anyone aged 15 years or more.
Arm/Group | Parent/Child With Children With Medical Complexity (CMC) | School Staff
Number analyzed (Participants) | 47 | 24
Number analyzed (BinaxNOW Rapid Antigen COVID-19 Tests) | 1403 | 965
Symptomatic BinaxNow Rapid Antigen Tests | 195 | 39

4. Primary Outcome: Change in Positive Rate: Number of Positive COVID-19 Tests Compared to Total Number of Tests Performed
Description: Data will be retrieved from study log.
Time Frame: Study duration (up to 21 months)
Measure: Number; unit: Positive BinaxNOW Rapid Antigen Tests
Units Other Than Participants: BinaxNOW Rapid Antigen COVID-19 Tests
Arm/Group | Parent/Child With Children With Medical Complexity (CMC) | School Staff
Number analyzed (Participants) | 47 | 24
Number analyzed (BinaxNOW Rapid Antigen COVID-19 Tests) | 1403 | 965
Positive BinaxNOW Rapid Antigen Tests | 30 | 5

5. Primary Outcome: Change in False-positive Rate: Number of Negative Confirmatory Polymerase Chain Reaction (PCR) as Compared to Total PCR Run for COVID-19 Testing
Description: Data will be retrieved from study log. All children and staff (n = 71) were included in this outcome. However, participants were not required to and were sometimes unable to complete a confirmatory PCR test after a positive in-home rapid test. This explains the difference between the number of positive at-home COVID-19 tests and the number of PCR tests.
  Some participants completed multiple confirmatory PCR tests over the study time frame. This explains why the PCR quantity is greater than the number of participants.
Time Frame: Study duration (up to 21 months)
Measure: Number; unit: Negative confirmatory PCRs
Units Other Than Participants: COVID-19 PCR Tests
Groups:
- Child With Children With Medical Complexity (CMC): 65 children and their parents will be recruited to participate. School staff will send a letter to all parents with children enrolled in the Waisman Early Childhood Program (WECP) inviting them to participate. Families new to the school or who initially decline participation and then reconsider may join at any time. Participants will also be offered the option of as needed symptomatic home testing.
  Additionally, parents who are vaccinated will be asked to participate in testing. Siblings may be enrolled in the study.
  BinaxNOW Rapid Antigen System: BinaxNOW Rapid Antigen System (Abbott) is a point-of-care, lateral flow immunoassay intended for the qualitative detection of nucleocapsid protein antigen from SARS-CoV-2 in direct anterior nasal (nares) swabs. Internal controls are built into the testing system and results are available in 15 minutes.
  The use of the BinaxNOW system is authorized under the Food and Drug Administration's Emergency Use Authorization. The test is allowed for over-the-counter, non-prescription use with or without symptoms. The test may be used with children two years and older with the help of sample collection by an adult, and the test may be self-administered by anyone aged 15 years or more.
Arm/Group | Child With Children With Medical Complexity (CMC) | School Staff
Number analyzed (Participants) | 27 | 8
Number analyzed (COVID-19 PCR Tests) | 49 | 15
Negative confirmatory PCRs | 22 | 1

6. Primary Outcome: Caregiver Change in Susceptibility: Number of Fully Vaccinated People Who Interact With Participant's Child at School
Description: * "How many of the people who interact with your child at school have been fully vaccinated?"
  * Response options: "None", "A few", "Some" "Most", "All", "Don't Know"
  * Dichotomized into: ("Most" or "All") vs. ("None", "A few", "Some", "Don't Know)
  * This question was only asked to caregivers.
  * Caregivers with multiple children enrolled completed a survey for each child.
Time Frame: Baseline, 3 month, 6 month, 9 month, 15 month, 18 month, 21 month, 24 month
Population: The number analyzed varies per row due to varied response rates per question at each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Parent/Child With Children With Medical Complexity (CMC)
Number analyzed (Participants) | 47
Participants
  Baseline: number analyzed (Participants) | 39
  Baseline: "Most" or "All" of the people who interact with their child at school have been fully vaccinated | 21
  Baseline: "None", "A few", "Some", "Don't Know" | 18
  3 month: number analyzed (Participants) | 29
  3 month: "Most" or "All" of the people who interact with their child at school have been fully vaccinated | 11
  3 month: "None", "A few", "Some", "Don't Know" | 18
  6 month: number analyzed (Participants) | 27
  6 month: "Most" or "All" of the people who interact with their child at school have been fully vaccinated | 15
  6 month: "None", "A few", "Some", "Don't Know" | 12
  9 month: number analyzed (Participants) | 18
  9 month: "Most" or "All" of the people who interact with their child at school have been fully vaccinated | 9
  9 month: "None", "A few", "Some", "Don't Know" | 9
  15 month: number analyzed (Participants) | 8
  15 month: "Most" or "All" of the people who interact with their child at school have been fully vaccinated | 4
  15 month: "None", "A few", "Some", "Don't Know" | 4
  18 month: number analyzed (Participants) | 8
  18 month: "Most" or "All" of the people who interact with their child at school have been fully vaccinated | 6
  18 month: "None", "A few", "Some", "Don't Know" | 2
  21 month: number analyzed (Participants) | 16
  21 month: "Most" or "All" of the people who interact with their child at school have been fully vaccinated | 7
  21 month: "None", "A few", "Some", "Don't Know" | 9
  24 month: number analyzed (Participants) | 10
  24 month: "Most" or "All" of the people who interact with their child at school have been fully vaccinated | 7
  24 month: "None", "A few", "Some", "Don't Know" | 3

7. Primary Outcome: Caregiver Change in Susceptibility: School Takes Precautions
Description: The following question from the Participant's perceived susceptibility survey will be answered dichotomously and presented qualitatively:
  * How comfortable are you with...the ability of your child's school to take all precautions to stop the spread of COVID-19?
  * Response options: "Not at all", "A little", "Somewhat", "Very", "Extremely"
  * Dichotomized into: ("Not at all", "A little", "Somewhat") vs. ("Very", "Extremely")
  * This question was only asked to caregivers.
  * Caregivers with multiple children enrolled completed a survey for each child.
Time Frame: Baseline, 3 month, 6 month, 9 month, 15 month, 18 month, 21 month, 24 month
Population: The number analyzed varies per row due to varied response rates per question at each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Parent/Child With Children With Medical Complexity (CMC)
Number analyzed (Participants) | 47
Participants
  Baseline: number analyzed (Participants) | 40
  Baseline: "Very" or "Extremely" comfortable | 27
  Baseline: "Not at all", "A little", or "Somewhat" comfortable | 13
  3 month: number analyzed (Participants) | 29
  3 month: "Very" or "Extremely" comfortable | 19
  3 month: "Not at all", "A little", or "Somewhat" comfortable | 10
  6 month: number analyzed (Participants) | 27
  6 month: "Very" or "Extremely" comfortable | 19
  6 month: "Not at all", "A little", or "Somewhat" comfortable | 8
  9 month: number analyzed (Participants) | 18
  9 month: "Very" or "Extremely" comfortable | 12
  9 month: "Not at all", "A little", or "Somewhat" comfortable | 6
  15 month: number analyzed (Participants) | 8
  15 month: "Very" or "Extremely" comfortable | 5
  15 month: "Not at all", "A little", or "Somewhat" comfortable | 3
  18 month: number analyzed (Participants) | 8
  18 month: "Very" or "Extremely" comfortable | 6
  18 month: "Not at all", "A little", or "Somewhat" comfortable | 2
  21 month: number analyzed (Participants) | 16
  21 month: "Very" or "Extremely" comfortable | 9
  21 month: "Not at all", "A little", or "Somewhat" comfortable | 7
  24 month: number analyzed (Participants) | 10
  24 month: "Very" or "Extremely" comfortable | 8
  24 month: "Not at all", "A little", or "Somewhat" comfortable | 2

8. Primary Outcome: Caregiver Change in Susceptibility: Likely to Get COVID-19
Description: Following questions from the Participant's perceived susceptibility survey will be answered dichotomously (agree or disagree) and presented qualitatively.
  * In your opinion, how likely is your child to get sick with COVID-19 by attending school in-person?
  * Response options: "Not at all", "A little", "Somewhat", "Very", "Extremely"
  * Dichotomized into: ("Not at all", "A little", "Somewhat") vs. ("Very", "Extremely")
  * This question was only asked to caregivers.
  * Caregivers with multiple children enrolled completed a survey for each child.
Time Frame: Baseline, 3 month, 6 month, 9 month, 15 month, 18 month, 21 month, 24 month
Population: The number analyzed varies per row due to varied response rates per question at each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Parent/Child With Children With Medical Complexity (CMC)
Number analyzed (Participants) | 47
Participants
  Baseline: number analyzed (Participants) | 39
  Baseline: "Very" or "Extremely" likely | 6
  Baseline: "Not at all", "A little", or "Somewhat" likely | 33
  3 month: number analyzed (Participants) | 29
  3 month: "Very" or "Extremely" likely | 5
  3 month: "Not at all", "A little", or "Somewhat" likely | 24
  6 month: number analyzed (Participants) | 28
  6 month: "Very" or "Extremely" likely | 3
  6 month: "Not at all", "A little", or "Somewhat" likely | 25
  9 month: number analyzed (Participants) | 18
  9 month: "Very" or "Extremely" likely | 3
  9 month: "Not at all", "A little", or "Somewhat" likely | 15
  15 month: number analyzed (Participants) | 8
  15 month: "Very" or "Extremely" likely | 2
  15 month: "Not at all", "A little", or "Somewhat" likely | 6
  18 month: number analyzed (Participants) | 8
  18 month: "Very" or "Extremely" likely | 2
  18 month: "Not at all", "A little", or "Somewhat" likely | 6
  21 month: number analyzed (Participants) | 16
  21 month: "Very" or "Extremely" likely | 7
  21 month: "Not at all", "A little", or "Somewhat" likely | 9
  24 month: number analyzed (Participants) | 10
  24 month: "Very" or "Extremely" likely | 1
  24 month: "Not at all", "A little", or "Somewhat" likely | 9

9. Primary Outcome: Change in Percentage of Caregivers for Perceived Severity Survey Question: Health Severely Affected
Description: Parent survey perceived severity construct variables will include:
  * If your child was sick with COVID-19, how likely would...their health be severely affected
  * Response options: "Not at all", "A little", "Somewhat", "Very", "Extremely"
  * Dichotomized into: ("Not at all", "A little", "Somewhat") vs. ("Very", "Extremely")
  * This question was only asked to caregivers.
  * Caregivers with multiple children enrolled completed a survey for each child.
Time Frame: 15 month, 18 month, 21 month, 24 month
Population: The number analyzed varies per row due to varied response rates per question at each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Parent/Child With Children With Medical Complexity (CMC)
Number analyzed (Participants) | 39
Participants
  15 month: number analyzed (Participants) | 8
  15 month: "Very" or "Extremely" likely | 1
  15 month: "Not at all", "A little", or "Somewhat" likely | 7
  18 month: number analyzed (Participants) | 8
  18 month: "Very" or "Extremely" likely | 1
  18 month: "Not at all", "A little", or "Somewhat" likely | 7
  21 month: number analyzed (Participants) | 13
  21 month: "Very" or "Extremely" likely | 0
  21 month: "Not at all", "A little", or "Somewhat" likely | 13
  24 month: number analyzed (Participants) | 10
  24 month: "Very" or "Extremely" likely | 0
  24 month: "Not at all", "A little", or "Somewhat" likely | 10

10. Primary Outcome: Change in Percentage of Caregivers to the Perceived Severity Survey Question: Health Permanently Reduced
Description: Parent survey perceived severity construct variables will be:
  * "If your child was sick with COVID-19, how likely would...their health be permanently reduced"
  * Response options: "Not at all", "A little", "Somewhat", "Very", "Extremely"
  * Dichotomized into: ("Not at all", "A little", "Somewhat") vs. ("Very", "Extremely")
  * This question was only asked to caregivers.
  * Caregivers with multiple children enrolled completed a survey for each child.
Time Frame: 15 month, 18 month, 21 month, 24 month
Population: The number analyzed varies per row due to varied response rates per question at each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Parent/Child With Children With Medical Complexity (CMC)
Number analyzed (Participants) | 39
Participants
  15 month: number analyzed (Participants) | 8
  15 month: "Very" or "Extremely" likely | 1
  15 month: "Not at all", "A little", or "Somewhat" likely | 7
  18 month: number analyzed (Participants) | 8
  18 month: "Very" or "Extremely" likely | 1
  18 month: "Not at all", "A little", or "Somewhat" likely | 7
  21 month: number analyzed (Participants) | 13
  21 month: "Very" or "Extremely" likely | 0
  21 month: "Not at all", "A little", or "Somewhat" likely | 13
  24 month: number analyzed (Participants) | 10
  24 month: "Very" or "Extremely" likely | 0
  24 month: "Not at all", "A little", or "Somewhat" likely | 10

11. Primary Outcome: Change in Percentage of Caregivers to the Perceived Severity Survey Question: Grave Health Consequences
Description: Parent survey perceived severity construct variables will be:
  * "If my child was sick with COVID-19, they would have grave health consequences."
  * Response options: "Not at all", "A little", "Somewhat", "Very", "Extremely"
  * Dichotomized into: ("Not at all", "A little", "Somewhat") vs. ("Very", "Extremely")
  * This question was only asked to caregivers.
  * Caregivers with multiple children enrolled completed a survey for each child.
Time Frame: 15 month, 18 month, 21 month, 24 month
Population: The number analyzed varies per row due to varied response rates per question at each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Parent/Child With Children With Medical Complexity (CMC)
Number analyzed (Participants) | 39
Participants
  15 month: number analyzed (Participants) | 8
  15 month: "Very" or "Extremely" likely | 1
  15 month: "Not at all", "A little", or "Somewhat" likely | 7
  18 month: number analyzed (Participants) | 8
  18 month: "Very" or "Extremely" likely | 1
  18 month: "Not at all", "A little", or "Somewhat" likely | 7
  21 month: number analyzed (Participants) | 13
  21 month: "Very" or "Extremely" likely | 0
  21 month: "Not at all", "A little", or "Somewhat" likely | 13
  24 month: number analyzed (Participants) | 10
  24 month: "Very" or "Extremely" likely | 0
  24 month: "Not at all", "A little", or "Somewhat" likely | 10

12. Primary Outcome: Caregiver Change in Motivation for Child to Attend School (Quite a Bit / a Great Deal vs Not)
Description: Participants will answer the following survey question in quite a bit / a great deal vs not:
  * "Based on the situation right now, how much do you want your child to attend school in-person at least some of the time?"
  * This question was only asked to caregivers.
  * Caregivers with multiple children enrolled completed a survey for each child.
Time Frame: Baseline, 3 month, 6 month, 9 month, 15 month, 18 month, 21 month, 24 month
Population: The number analyzed varies per row due to varied response rates per question at each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Parent/Child With Children With Medical Complexity (CMC)
Number analyzed (Participants) | 47
Participants
  Baseline: number analyzed (Participants) | 39
  Baseline: "Quite a bit" or "A great deal" | 30
  Baseline: "Somewhat," "A little," or "Not at all" | 9
  3 month: number analyzed (Participants) | 30
  3 month: "Quite a bit" or "A great deal" | 26
  3 month: "Somewhat," "A little," or "Not at all" | 4
  6 month: number analyzed (Participants) | 27
  6 month: "Quite a bit" or "A great deal" | 26
  6 month: "Somewhat," "A little," or "Not at all" | 1
  9 month: number analyzed (Participants) | 18
  9 month: "Quite a bit" or "A great deal" | 15
  9 month: "Somewhat," "A little," or "Not at all" | 3
  15 month: number analyzed (Participants) | 8
  15 month: "Quite a bit" or "A great deal" | 8
  15 month: "Somewhat," "A little," or "Not at all" | 0
  18 month: number analyzed (Participants) | 8
  18 month: "Quite a bit" or "A great deal" | 8
  18 month: "Somewhat," "A little," or "Not at all" | 0
  21 month: number analyzed (Participants) | 16
  21 month: "Quite a bit" or "A great deal" | 16
  21 month: "Somewhat," "A little," or "Not at all" | 0
  24 month: number analyzed (Participants) | 10
  24 month: "Quite a bit" or "A great deal" | 10
  24 month: "Somewhat," "A little," or "Not at all" | 0

13. Primary Outcome: Caregiver Change in Perceived Benefits to Child Attending School: Important to Health
Description: Parent survey perceived benefits construct survey will be having 6 questions ranging from benefits to child's overall health, therapy needs, impact on family. Survey will be analyzed qualitatively.
  * How important is attending school in-person to your child's overall health?
  * Dichotomized into: ("Not at all important", "A little important", "Somewhat important") vs. ("Very important", "Extremely important")
  * This question was only asked to caregivers.
  * Caregivers with multiple children enrolled completed a survey for each child.
Time Frame: Baseline, 3 month, 6 month, 9 month, 15 month, 18 month, 21 month, 24 month
Population: The number analyzed varies per row due to varied response rates per question at each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Parent/Child With Children With Medical Complexity (CMC)
Number analyzed (Participants) | 47
Participants
  Baseline: number analyzed (Participants) | 40
  Baseline: "Very important" or "Extremely important" | 32
  Baseline: "Not at all important", "A little important", or "Somewhat important" | 8
  3 month: number analyzed (Participants) | 30
  3 month: "Very important" or "Extremely important" | 21
  3 month: "Not at all important", "A little important", or "Somewhat important" | 9
  6 month: number analyzed (Participants) | 28
  6 month: "Very important" or "Extremely important" | 21
  6 month: "Not at all important", "A little important", or "Somewhat important" | 7
  9 month: number analyzed (Participants) | 18
  9 month: "Very important" or "Extremely important" | 15
  9 month: "Not at all important", "A little important", or "Somewhat important" | 3
  15 month: number analyzed (Participants) | 8
  15 month: "Very important" or "Extremely important" | 8
  15 month: "Not at all important", "A little important", or "Somewhat important" | 0
  18 month: number analyzed (Participants) | 8
  18 month: "Very important" or "Extremely important" | 7
  18 month: "Not at all important", "A little important", or "Somewhat important" | 1
  21 month: number analyzed (Participants) | 16
  21 month: "Very important" or "Extremely important" | 13
  21 month: "Not at all important", "A little important", or "Somewhat important" | 3
  24 month: number analyzed (Participants) | 10
  24 month: "Very important" or "Extremely important" | 9
  24 month: "Not at all important", "A little important", or "Somewhat important" | 1

14. Primary Outcome: Caregiver Change in Perceived Benefits to Child Attending School: In-person Schooling
Description: Parent survey perceived benefits construct survey will be having 6 questions ranging from benefits to child's overall health, therapy needs, and impact on family. Survey will be analyzed qualitatively.
  * Compared to fully virtual school, how much better or worse is attending any school in-person for your child?
  * Dichotomized into: ("Quite a bit worse", "Somewhat worse", "A little bit worse", "Neither better nor worse") vs. ("A little bit better", "Somewhat better", "Quite a bit better")
  * This question was only asked to caregivers.
  * Caregivers with multiple children enrolled completed a survey for each child.
Time Frame: Baseline, 3 month, 6 month, 9 month, 15 month, 18 month, 21 month, 24 month
Population: The number analyzed varies per row due to varied response rates per question at each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Parent/Child With Children With Medical Complexity (CMC)
Number analyzed (Participants) | 47
Participants
  Baseline: number analyzed (Participants) | 38
  Baseline: "A little bit better", "Somewhat better", or "Quite a bit better" | 36
  Baseline: "Quite a bit worse", "Somewhat worse", "A little bit worse", or "Neither better nor worse" | 2
  3 month: number analyzed (Participants) | 29
  3 month: "A little bit better", "Somewhat better", or "Quite a bit better" | 27
  3 month: "Quite a bit worse", "Somewhat worse", "A little bit worse", or "Neither better nor worse" | 2
  6 month: number analyzed (Participants) | 28
  6 month: "A little bit better", "Somewhat better", or "Quite a bit better" | 26
  6 month: "Quite a bit worse", "Somewhat worse", "A little bit worse", or "Neither better nor worse" | 2
  9 month: number analyzed (Participants) | 18
  9 month: "A little bit better", "Somewhat better", or "Quite a bit better" | 16
  9 month: "Quite a bit worse", "Somewhat worse", "A little bit worse", or "Neither better nor worse" | 2
  15 month: number analyzed (Participants) | 8
  15 month: "A little bit better", "Somewhat better", or "Quite a bit better" | 8
  15 month: "Quite a bit worse", "Somewhat worse", "A little bit worse", or "Neither better nor worse" | 0
  18 month: number analyzed (Participants) | 8
  18 month: "A little bit better", "Somewhat better", or "Quite a bit better" | 7
  18 month: "Quite a bit worse", "Somewhat worse", "A little bit worse", or "Neither better nor worse" | 1
  21 month: number analyzed (Participants) | 15
  21 month: "A little bit better", "Somewhat better", or "Quite a bit better" | 15
  21 month: "Quite a bit worse", "Somewhat worse", "A little bit worse", or "Neither better nor worse" | 0
  24 month: number analyzed (Participants) | 8
  24 month: "A little bit better", "Somewhat better", or "Quite a bit better" | 8
  24 month: "Quite a bit worse", "Somewhat worse", "A little bit worse", or "Neither better nor worse" | 0

15. Primary Outcome: Caregiver Change in Perceived Benefits to Child Attending School: Therapy Needs
Description: Parent survey perceived benefits construct survey will be having 6 questions ranging from benefits to child's overall health, therapy needs, impact on family. Survey will be analyzed qualitatively.
  * How much of your child's therapy needs are only met by attending school in-person?
  * Dichotomized into: ("None", "A few", "Some" vs. "Most", "All")
  * This question was only asked to caregivers.
  * Caregivers with multiple children enrolled completed a survey for each child.
Time Frame: Baseline, 3 month, 6 month, 9 month, 15 month, 18 month, 21 month, 24 month
Population: The number analyzed varies per row due to varied response rates per question at each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Parent/Child With Children With Medical Complexity (CMC)
Number analyzed (Participants) | 47
Participants
  Baseline: number analyzed (Participants) | 31
  Baseline: "Most", "All" | 9
  Baseline: "None", "A few", "Some" | 22
  3 month: number analyzed (Participants) | 23
  3 month: "Most", "All" | 9
  3 month: "None", "A few", "Some" | 14
  6 month: number analyzed (Participants) | 20
  6 month: "Most", "All" | 10
  6 month: "None", "A few", "Some" | 10
  9 month: number analyzed (Participants) | 16
  9 month: "Most", "All" | 8
  9 month: "None", "A few", "Some" | 8
  15 month: number analyzed (Participants) | 5
  15 month: "Most", "All" | 2
  15 month: "None", "A few", "Some" | 3
  18 month: number analyzed (Participants) | 6
  18 month: "Most", "All" | 2
  18 month: "None", "A few", "Some" | 4
  21 month: number analyzed (Participants) | 11
  21 month: "Most", "All" | 4
  21 month: "None", "A few", "Some" | 7
  24 month: number analyzed (Participants) | 8
  24 month: "Most", "All" | 2
  24 month: "None", "A few", "Some" | 6

16. Primary Outcome: Caregiver Change in Perceived Benefits to Child Attending School: Positive for Family
Description: Parent survey perceived benefits construct survey will be having 6 questions ranging from benefits to child's overall health, therapy needs, impact on family. Survey will be analyzed qualitatively.
  * How positive or negative is your child attending school in-person for...your family
  * Dichotomized into: ("Very negative", "Somewhat negative", "A little negative", "Neutral") vs. ("A little positive", "Somewhat positive", "Very positive")
  * This question was only asked to caregivers.
  * Caregivers with multiple children enrolled completed a survey for each child.
Time Frame: Baseline, 3 month, 6 month, 9 month, 15 month, 18 month, 21 month, 24 month
Population: The number analyzed varies per row due to varied response rates per question at each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Parent/Child With Children With Medical Complexity (CMC)
Number analyzed (Participants) | 47
Participants
  Baseline: number analyzed (Participants) | 40
  Baseline: "A little positive", "Somewhat positive", or "Very positive" | 39
  Baseline: "Very negative", "Somewhat negative", or "A little negative", "Neutral" | 1
  3 month: number analyzed (Participants) | 29
  3 month: "A little positive", "Somewhat positive", or "Very positive" | 29
  3 month: "Very negative", "Somewhat negative", or "A little negative", "Neutral" | 0
  6 month: number analyzed (Participants) | 28
  6 month: "A little positive", "Somewhat positive", or "Very positive" | 27
  6 month: "Very negative", "Somewhat negative", or "A little negative", "Neutral" | 1
  9 month: number analyzed (Participants) | 18
  9 month: "A little positive", "Somewhat positive", or "Very positive" | 18
  9 month: "Very negative", "Somewhat negative", or "A little negative", "Neutral" | 0
  15 month: number analyzed (Participants) | 8
  15 month: "A little positive", "Somewhat positive", or "Very positive" | 8
  15 month: "Very negative", "Somewhat negative", or "A little negative", "Neutral" | 0
  18 month: number analyzed (Participants) | 8
  18 month: "A little positive", "Somewhat positive", or "Very positive" | 8
  18 month: "Very negative", "Somewhat negative", or "A little negative", "Neutral" | 0
  21 month: number analyzed (Participants) | 16
  21 month: "A little positive", "Somewhat positive", or "Very positive" | 16
  21 month: "Very negative", "Somewhat negative", or "A little negative", "Neutral" | 0
  24 month: number analyzed (Participants) | 10
  24 month: "A little positive", "Somewhat positive", or "Very positive" | 10
  24 month: "Very negative", "Somewhat negative", or "A little negative", "Neutral" | 0

17. Primary Outcome: Caregiver Change in Perceived Benefits to Child Attending School: Positive for Staff
Description: Parent survey perceived benefits construct survey will be having 6 questions ranging from benefits to child's overall health, therapy needs, impact on family. Survey will be analyzed qualitatively.
  * How positive or negative is your child attending school in-person for...the staff and teachers
  * Dichotomized into: ("Very negative", "Somewhat negative", "A little negative", "Neutral") vs. ("A little positive", "Somewhat positive", "Very positive")
  * This question was only asked to caregivers.
  * Caregivers with multiple children enrolled completed a survey for each child.
Time Frame: Baseline, 3 month, 6 month, 9 month, 15 month, 18 month, 21 month, 24 month
Population: The number analyzed varies per row due to varied response rates per question at each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Parent/Child With Children With Medical Complexity (CMC)
Number analyzed (Participants) | 47
Participants
  Baseline: number analyzed (Participants) | 40
  Baseline: "A little positive", "Somewhat positive", or "Very positive" | 32
  Baseline: "Very negative", "Somewhat negative", or "A little negative", "Neutral" | 8
  3 month: number analyzed (Participants) | 29
  3 month: "A little positive", "Somewhat positive", or "Very positive" | 23
  3 month: "Very negative", "Somewhat negative", or "A little negative", "Neutral" | 6
  6 month: number analyzed (Participants) | 28
  6 month: "A little positive", "Somewhat positive", or "Very positive" | 22
  6 month: "Very negative", "Somewhat negative", or "A little negative", "Neutral" | 6
  9 month: number analyzed (Participants) | 17
  9 month: "A little positive", "Somewhat positive", or "Very positive" | 15
  9 month: "Very negative", "Somewhat negative", or "A little negative", "Neutral" | 2
  15 month: number analyzed (Participants) | 8
  15 month: "A little positive", "Somewhat positive", or "Very positive" | 7
  15 month: "Very negative", "Somewhat negative", or "A little negative", "Neutral" | 1
  18 month: number analyzed (Participants) | 8
  18 month: "A little positive", "Somewhat positive", or "Very positive" | 6
  18 month: "Very negative", "Somewhat negative", or "A little negative", "Neutral" | 2
  21 month: number analyzed (Participants) | 15
  21 month: "A little positive", "Somewhat positive", or "Very positive" | 12
  21 month: "Very negative", "Somewhat negative", or "A little negative", "Neutral" | 3
  24 month: number analyzed (Participants) | 10
  24 month: "A little positive", "Somewhat positive", or "Very positive" | 10
  24 month: "Very negative", "Somewhat negative", or "A little negative", "Neutral" | 0

18. Primary Outcome: Caregiver Change in Perceived Benefits to Child Attending School: Keep Jobs
Description: Parent survey perceived benefits construct survey will be having 6 questions ranging from benefits to child's overall health, therapy needs, impact on family. Survey will be analyzed qualitatively.
  * Does your child attending school in-person help the adults in your family to keep their jobs?
  * Response options: Yes / No
  * This question was only asked to caregivers.
  * Caregivers with multiple children enrolled completed a survey for each child.
Time Frame: Baseline, 3 month, 6 month, 9 month, 15 month, 18 month, 21 month, 24 month
Population: The number analyzed varies per row due to varied response rates per question at each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Parent/Child With Children With Medical Complexity (CMC)
Number analyzed (Participants) | 47
Participants
  Baseline: number analyzed (Participants) | 39
  Baseline: Yes | 31
  Baseline: No | 8
  3 month: number analyzed (Participants) | 29
  3 month: Yes | 24
  3 month: No | 5
  6 month: number analyzed (Participants) | 28
  6 month: Yes | 23
  6 month: No | 5
  9 month: number analyzed (Participants) | 18
  9 month: Yes | 13
  9 month: No | 5
  15 month: number analyzed (Participants) | 8
  15 month: Yes | 7
  15 month: No | 1
  18 month: number analyzed (Participants) | 7
  18 month: Yes | 7
  18 month: No | 0
  21 month: number analyzed (Participants) | 16
  21 month: Yes | 14
  21 month: No | 2
  24 month: number analyzed (Participants) | 10
  24 month: Yes | 8
  24 month: No | 2

19. Primary Outcome: Caregiver Change in Barriers to School Attendance: Number of People
Description: Survey will have following questions which will be answered dichotomously very/extremely [comfortable] vs not.
  * How comfortable are you with the number of people around your child at school?
  * Dichotomized into: ("Not at all", "A little", "Somewhat") vs. ("Very", "Extremely")
  * This question was only asked to caregivers.
  * Caregivers with multiple children enrolled completed a survey for each child.
Time Frame: Baseline, 3 month, 6 month, 9 month, 15 month, 18 month, 21 month, 24 month
Population: The number analyzed varies per row due to varied response rates per question at each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Parent/Child With Children With Medical Complexity (CMC)
Number analyzed (Participants) | 47
Participants
  Baseline: number analyzed (Participants) | 40
  Baseline: "Very" or "Extremely" comfortable | 21
  Baseline: "Not at all", "A little", or "Somewhat" comfortable | 19
  3 month: number analyzed (Participants) | 29
  3 month: "Very" or "Extremely" comfortable | 10
  3 month: "Not at all", "A little", or "Somewhat" comfortable | 19
  6 month: number analyzed (Participants) | 27
  6 month: "Very" or "Extremely" comfortable | 15
  6 month: "Not at all", "A little", or "Somewhat" comfortable | 12
  9 month: number analyzed (Participants) | 17
  9 month: "Very" or "Extremely" comfortable | 11
  9 month: "Not at all", "A little", or "Somewhat" comfortable | 6
  15 month: number analyzed (Participants) | 8
  15 month: "Very" or "Extremely" comfortable | 4
  15 month: "Not at all", "A little", or "Somewhat" comfortable | 4
  18 month: number analyzed (Participants) | 8
  18 month: "Very" or "Extremely" comfortable | 5
  18 month: "Not at all", "A little", or "Somewhat" comfortable | 3
  21 month: number analyzed (Participants) | 16
  21 month: "Very" or "Extremely" comfortable | 12
  21 month: "Not at all", "A little", or "Somewhat" comfortable | 4
  24 month: number analyzed (Participants) | 10
  24 month: "Very" or "Extremely" comfortable | 7
  24 month: "Not at all", "A little", or "Somewhat" comfortable | 3

20. Primary Outcome: Caregiver Change in Barriers to School Attendance: Proximity
Description: Survey will have following questions which will be answered dichotomously very/extremely [comfortable] vs not.
  * How comfortable are you with how close people have to be to your child at school?
  * Dichotomized into: ("Not at all", "A little", "Somewhat") vs. ("Very", "Extremely")
  * This question was only asked to caregivers.
  * Caregivers with multiple children enrolled completed a survey for each child.
Time Frame: Baseline, 3 month, 6 month, 9 month, 15 month, 18 month, 21 month, 24 month
Population: The number analyzed varies per row due to varied response rates per question at each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Parent/Child With Children With Medical Complexity (CMC)
Number analyzed (Participants) | 47
Participants
  Baseline: number analyzed (Participants) | 40
  Baseline: "Very" or "Extremely" comfortable | 20
  Baseline: "Not at all", "A little", or "Somewhat" comfortable | 20
  3 month: number analyzed (Participants) | 29
  3 month: "Very" or "Extremely" comfortable | 9
  3 month: "Not at all", "A little", or "Somewhat" comfortable | 20
  6 month: number analyzed (Participants) | 27
  6 month: "Very" or "Extremely" comfortable | 13
  6 month: "Not at all", "A little", or "Somewhat" comfortable | 14
  9 month: number analyzed (Participants) | 18
  9 month: "Very" or "Extremely" comfortable | 10
  9 month: "Not at all", "A little", or "Somewhat" comfortable | 8
  15 month: number analyzed (Participants) | 8
  15 month: "Very" or "Extremely" comfortable | 4
  15 month: "Not at all", "A little", or "Somewhat" comfortable | 4
  18 month: number analyzed (Participants) | 8
  18 month: "Very" or "Extremely" comfortable | 3
  18 month: "Not at all", "A little", or "Somewhat" comfortable | 5
  21 month: number analyzed (Participants) | 15
  21 month: "Very" or "Extremely" comfortable | 10
  21 month: "Not at all", "A little", or "Somewhat" comfortable | 5
  24 month: number analyzed (Participants) | 10
  24 month: "Very" or "Extremely" comfortable | 6
  24 month: "Not at all", "A little", or "Somewhat" comfortable | 4

21. Primary Outcome: Caregiver Change in Barriers to School Attendance: PPE
Description: Survey will have following questions which will be answered dichotomously very/extremely [comfortable] vs not.
  * How comfortable are you with the amount personal protective equipment (PPE), such as masks and gloves, available at school?
  * Dichotomized into: ("Not at all", "A little", "Somewhat") vs. ("Very", "Extremely")
  * This question was only asked to caregivers.
  * Caregivers with multiple children enrolled completed a survey for each child.
Time Frame: Baseline, 3 month, 6 month, 9 month, 15 month, 18 month, 21 month, 24 month
Population: The number analyzed varies per row due to varied response rates per question at each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Parent/Child With Children With Medical Complexity (CMC)
Number analyzed (Participants) | 47
Participants
  Baseline: number analyzed (Participants) | 40
  Baseline: "Very" or "Extremely" comfortable | 27
  Baseline: "Not at all", "A little", or "Somewhat" comfortable | 13
  3 month: number analyzed (Participants) | 29
  3 month: "Very" or "Extremely" comfortable | 16
  3 month: "Not at all", "A little", or "Somewhat" comfortable | 13
  6 month: number analyzed (Participants) | 26
  6 month: "Very" or "Extremely" comfortable | 16
  6 month: "Not at all", "A little", or "Somewhat" comfortable | 10
  9 month: number analyzed (Participants) | 18
  9 month: "Very" or "Extremely" comfortable | 17
  9 month: "Not at all", "A little", or "Somewhat" comfortable | 1
  15 month: number analyzed (Participants) | 8
  15 month: "Very" or "Extremely" comfortable | 3
  15 month: "Not at all", "A little", or "Somewhat" comfortable | 5
  18 month: number analyzed (Participants) | 8
  18 month: "Very" or "Extremely" comfortable | 5
  18 month: "Not at all", "A little", or "Somewhat" comfortable | 3
  21 month: number analyzed (Participants) | 16
  21 month: "Very" or "Extremely" comfortable | 11
  21 month: "Not at all", "A little", or "Somewhat" comfortable | 5
  24 month: number analyzed (Participants) | 10
  24 month: "Very" or "Extremely" comfortable | 7
  24 month: "Not at all", "A little", or "Somewhat" comfortable | 3

22. Primary Outcome: Caregiver Change in Barriers to School Attendance: Testing
Description: Survey will have following questions which will be answered dichotomously very/extremely [comfortable] vs not.
  * How comfortable are you with the amount of COVID-19 testing among school staff and classmates?
  * Dichotomized into: ("Not at all", "A little", "Somewhat") vs. ("Very", "Extremely")
  * This question was only asked to caregivers.
  * Caregivers with multiple children enrolled completed a survey for each child.
Time Frame: Baseline, 3 month, 6 month, 9 month, 15 month, 18 month, 21 month, 24 month
Population: The number analyzed varies per row due to varied response rates per question at each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Parent/Child With Children With Medical Complexity (CMC)
Number analyzed (Participants) | 47
Participants
  Baseline: number analyzed (Participants) | 40
  Baseline: "Very" or "Extremely" comfortable | 30
  Baseline: "Not at all", "A little", or "Somewhat" comfortable | 10
  3 month: number analyzed (Participants) | 29
  3 month: "Very" or "Extremely" comfortable | 19
  3 month: "Not at all", "A little", or "Somewhat" comfortable | 10
  6 month: number analyzed (Participants) | 26
  6 month: "Very" or "Extremely" comfortable | 13
  6 month: "Not at all", "A little", or "Somewhat" comfortable | 13
  9 month: number analyzed (Participants) | 18
  9 month: "Very" or "Extremely" comfortable | 11
  9 month: "Not at all", "A little", or "Somewhat" comfortable | 7
  15 month: number analyzed (Participants) | 8
  15 month: "Very" or "Extremely" comfortable | 3
  15 month: "Not at all", "A little", or "Somewhat" comfortable | 5
  18 month: number analyzed (Participants) | 8
  18 month: "Very" or "Extremely" comfortable | 5
  18 month: "Not at all", "A little", or "Somewhat" comfortable | 3
  21 month: number analyzed (Participants) | 16
  21 month: "Very" or "Extremely" comfortable | 12
  21 month: "Not at all", "A little", or "Somewhat" comfortable | 4
  24 month: number analyzed (Participants) | 10
  24 month: "Very" or "Extremely" comfortable | 8
  24 month: "Not at all", "A little", or "Somewhat" comfortable | 2

23. Primary Outcome: Caregiver Change in Barriers to School Attendance: Following Recommendations
Description: Survey will have following questions which will be answered dichotomously very/extremely [comfortable] vs not.
  * How comfortable are you with how closely parents of classmates follow recommendations to keep your child safe?
  * Dichotomized into: ("Not at all", "A little", "Somewhat") vs. ("Very", "Extremely")
  * This question was only asked to caregivers.
  * Caregivers with multiple children enrolled completed a survey for each child.
Time Frame: Baseline, 3 month, 6 month, 9 month, 15 month, 18 month, 21 month, 24 month
Population: The number analyzed varies per row due to varied response rates per question at each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Parent/Child With Children With Medical Complexity (CMC)
Number analyzed (Participants) | 47
Participants
  Baseline: number analyzed (Participants) | 40
  Baseline: "Very" or "Extremely" comfortable | 23
  Baseline: "Not at all", "A little", or "Somewhat" comfortable | 17
  3 month: number analyzed (Participants) | 29
  3 month: "Very" or "Extremely" comfortable | 10
  3 month: "Not at all", "A little", or "Somewhat" comfortable | 19
  6 month: number analyzed (Participants) | 26
  6 month: "Very" or "Extremely" comfortable | 14
  6 month: "Not at all", "A little", or "Somewhat" comfortable | 12
  9 month: number analyzed (Participants) | 16
  9 month: "Very" or "Extremely" comfortable | 14
  9 month: "Not at all", "A little", or "Somewhat" comfortable | 2
  15 month: number analyzed (Participants) | 8
  15 month: "Very" or "Extremely" comfortable | 4
  15 month: "Not at all", "A little", or "Somewhat" comfortable | 4
  18 month: number analyzed (Participants) | 8
  18 month: "Very" or "Extremely" comfortable | 5
  18 month: "Not at all", "A little", or "Somewhat" comfortable | 3
  21 month: number analyzed (Participants) | 15
  21 month: "Very" or "Extremely" comfortable | 11
  21 month: "Not at all", "A little", or "Somewhat" comfortable | 4
  24 month: number analyzed (Participants) | 10
  24 month: "Very" or "Extremely" comfortable | 7
  24 month: "Not at all", "A little", or "Somewhat" comfortable | 3

24. Primary Outcome: Caregiver Change in Barriers to School Attendance: Transportation
Description: Survey will have following questions which will be answered dichotomously very/extremely vs not.
  * How difficult is it to transport your child to or from school as a result of COVID-19?
  * Dichotomized as: ("Not at all", "A little", "Somewhat") vs. ("Very", "Extremely")
  * This question was only asked to caregivers.
  * Caregivers with multiple children enrolled completed a survey for each child.
Time Frame: Baseline, 3 month, 6 month, 9 month, 15 month, 18 month, 21 month, 24 month
Population: The number analyzed varies per row due to varied response rates per question at each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Parent/Child With Children With Medical Complexity (CMC)
Number analyzed (Participants) | 47
Participants
  Baseline: number analyzed (Participants) | 40
  Baseline: "Very" or "Extremely" difficult | 1
  Baseline: "Not at all", "A little", or "Somewhat" difficult | 39
  3 month: number analyzed (Participants) | 29
  3 month: "Very" or "Extremely" difficult | 0
  3 month: "Not at all", "A little", or "Somewhat" difficult | 29
  6 month: number analyzed (Participants) | 28
  6 month: "Very" or "Extremely" difficult | 1
  6 month: "Not at all", "A little", or "Somewhat" difficult | 27
  9 month: number analyzed (Participants) | 18
  9 month: "Very" or "Extremely" difficult | 1
  9 month: "Not at all", "A little", or "Somewhat" difficult | 17
  15 month: number analyzed (Participants) | 8
  15 month: "Very" or "Extremely" difficult | 0
  15 month: "Not at all", "A little", or "Somewhat" difficult | 8
  18 month: number analyzed (Participants) | 8
  18 month: "Very" or "Extremely" difficult | 0
  18 month: "Not at all", "A little", or "Somewhat" difficult | 8
  21 month: number analyzed (Participants) | 16
  21 month: "Very" or "Extremely" difficult | 0
  21 month: "Not at all", "A little", or "Somewhat" difficult | 16
  24 month: number analyzed (Participants) | 10
  24 month: "Very" or "Extremely" difficult | 0
  24 month: "Not at all", "A little", or "Somewhat" difficult | 10

25. Primary Outcome: Caregiver Change in Barriers to School Attendance: Wash
Description: Survey will have following questions which will be answered dichotomously very/extremely vs not.
  * In your child's school, do they have access to necessary facilities to wash?
  * Dichotomized as: ("Yes, all of the time", "Yes, most of the time") vs. ("Some of the time", "Rarely", "Not at all")
  * This question was only asked to caregivers.
  * Caregivers with multiple children enrolled completed a survey for each child.
Time Frame: Baseline, 3 month, 6 month, 9 month, 15 month, 18 month, 21 month, 24 month
Population: The number analyzed varies per row due to varied response rates per question at each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Parent/Child With Children With Medical Complexity (CMC)
Number analyzed (Participants) | 47
Participants
  Baseline: number analyzed (Participants) | 39
  Baseline: "Yes, all of the time" or "Yes, most of the time" | 39
  Baseline: "Some of the time", "Rarely", or "Not at all" | 0
  3 month: number analyzed (Participants) | 29
  3 month: "Yes, all of the time" or "Yes, most of the time" | 29
  3 month: "Some of the time", "Rarely", or "Not at all" | 0
  6 month: number analyzed (Participants) | 28
  6 month: "Yes, all of the time" or "Yes, most of the time" | 28
  6 month: "Some of the time", "Rarely", or "Not at all" | 0
  9 month: number analyzed (Participants) | 18
  9 month: "Yes, all of the time" or "Yes, most of the time" | 18
  9 month: "Some of the time", "Rarely", or "Not at all" | 0
  15 month: number analyzed (Participants) | 8
  15 month: "Yes, all of the time" or "Yes, most of the time" | 8
  15 month: "Some of the time", "Rarely", or "Not at all" | 0
  18 month: number analyzed (Participants) | 8
  18 month: "Yes, all of the time" or "Yes, most of the time" | 8
  18 month: "Some of the time", "Rarely", or "Not at all" | 0
  21 month: number analyzed (Participants) | 16
  21 month: "Yes, all of the time" or "Yes, most of the time" | 16
  21 month: "Some of the time", "Rarely", or "Not at all" | 0
  24 month: number analyzed (Participants) | 10
  24 month: "Yes, all of the time" or "Yes, most of the time" | 10
  24 month: "Some of the time", "Rarely", or "Not at all" | 0

26. Primary Outcome: Caregiver Change in Barriers to School Attendance: Close Contact
Description: Survey will have following questions which will be answered dichotomously very/extremely [comfortable] vs not.
  * While in school, is your child required to be in close contact (i.e., within 6 ft) with others? 'Others' includes teachers, aides, nurses, and classmates.
  * Dichotomized as: ("Yes, all of the time", "Yes, most of the time") vs. ("Some of the time", "Rarely", "Not at all")
  * This question was only asked to caregivers.
  * Caregivers with multiple children enrolled completed a survey for each child.
Time Frame: Baseline, 3 month, 6 month, 9 month, 15 month, 18 month, 21 month, 24 month
Population: The number analyzed varies per row due to varied response rates per question at each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Parent/Child With Children With Medical Complexity (CMC)
Number analyzed (Participants) | 47
Participants
  Baseline: number analyzed (Participants) | 40
  Baseline: "Yes, all of the time" or "Yes, most of the time" | 24
  Baseline: "Some of the time", "Rarely", or "Not at all" | 16
  3 month: number analyzed (Participants) | 29
  3 month: "Yes, all of the time" or "Yes, most of the time" | 21
  3 month: "Some of the time", "Rarely", or "Not at all" | 8
  6 month: number analyzed (Participants) | 28
  6 month: "Yes, all of the time" or "Yes, most of the time" | 24
  6 month: "Some of the time", "Rarely", or "Not at all" | 4
  9 month: number analyzed (Participants) | 18
  9 month: "Yes, all of the time" or "Yes, most of the time" | 15
  9 month: "Some of the time", "Rarely", or "Not at all" | 3
  15 month: number analyzed (Participants) | 8
  15 month: "Yes, all of the time" or "Yes, most of the time" | 6
  15 month: "Some of the time", "Rarely", or "Not at all" | 2
  18 month: number analyzed (Participants) | 8
  18 month: "Yes, all of the time" or "Yes, most of the time" | 6
  18 month: "Some of the time", "Rarely", or "Not at all" | 2
  21 month: number analyzed (Participants) | 15
  21 month: "Yes, all of the time" or "Yes, most of the time" | 13
  21 month: "Some of the time", "Rarely", or "Not at all" | 2
  24 month: number analyzed (Participants) | 10
  24 month: "Yes, all of the time" or "Yes, most of the time" | 8
  24 month: "Some of the time", "Rarely", or "Not at all" | 2

27. Primary Outcome: Caregiver Change in Barriers to School Attendance: Masking
Description: Survey will have following questions which will be answered dichotomously very/extremely vs not.
  * While in school, is your child able to wear a mask?
  * Dichotomized as: ("Yes, all of the time", "Yes, most of the time") vs. ("Some of the time", "Rarely", "Not at all")
  * This question was only asked to caregivers.
  * Caregivers with multiple children enrolled completed a survey for each child.
Time Frame: Baseline, 3 month, 6 month, 9 month, 15 month, 18 month, 21 month, 24 month
Population: The number analyzed varies per row due to varied response rates per question at each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Parent/Child With Children With Medical Complexity (CMC)
Number analyzed (Participants) | 47
Participants
  Baseline: number analyzed (Participants) | 40
  Baseline: "Yes, all of the time" or "Yes, most of the time" | 30
  Baseline: "Some of the time", "Rarely", or "Not at all" | 10
  3 month: number analyzed (Participants) | 29
  3 month: "Yes, all of the time" or "Yes, most of the time" | 23
  3 month: "Some of the time", "Rarely", or "Not at all" | 6
  6 month: number analyzed (Participants) | 28
  6 month: "Yes, all of the time" or "Yes, most of the time" | 23
  6 month: "Some of the time", "Rarely", or "Not at all" | 5
  9 month: number analyzed (Participants) | 18
  9 month: "Yes, all of the time" or "Yes, most of the time" | 14
  9 month: "Some of the time", "Rarely", or "Not at all" | 4
  15 month: number analyzed (Participants) | 8
  15 month: "Yes, all of the time" or "Yes, most of the time" | 3
  15 month: "Some of the time", "Rarely", or "Not at all" | 5
  18 month: number analyzed (Participants) | 8
  18 month: "Yes, all of the time" or "Yes, most of the time" | 6
  18 month: "Some of the time", "Rarely", or "Not at all" | 2
  21 month: number analyzed (Participants) | 16
  21 month: "Yes, all of the time" or "Yes, most of the time" | 7
  21 month: "Some of the time", "Rarely", or "Not at all" | 9
  24 month: number analyzed (Participants) | 10
  24 month: "Yes, all of the time" or "Yes, most of the time" | 5
  24 month: "Some of the time", "Rarely", or "Not at all" | 5

28. Primary Outcome: Caregiver Change in Cues: Has a Teacher or Staff Member Encouraged Child to Attend School In-person? (Y/N)
Description: Participants will answer the following survey question in Yes/No:
  * "Teachers/staff have asked for my child to attend school."- Y/N
  * This question was only asked to caregivers.
  * Caregivers with multiple children enrolled completed a survey for each child.
Time Frame: Baseline, 3 month, 6 month, 9 month, 15 month, 18 month, 21 month, 24 month
Population: The number analyzed varies per row due to varied response rates per question at each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Parent/Child With Children With Medical Complexity (CMC)
Number analyzed (Participants) | 47
Participants
  Baseline: number analyzed (Participants) | 38
  Baseline: Yes | 7
  Baseline: No | 31
  3 month: number analyzed (Participants) | 29
  3 month: Yes | 7
  3 month: No | 22
  6 month: number analyzed (Participants) | 27
  6 month: Yes | 7
  6 month: No | 20
  9 month: number analyzed (Participants) | 18
  9 month: Yes | 6
  9 month: No | 12
  15 month: number analyzed (Participants) | 8
  15 month: Yes | 4
  15 month: No | 4
  18 month: number analyzed (Participants) | 8
  18 month: Yes | 3
  18 month: No | 5
  21 month: number analyzed (Participants) | 15
  21 month: Yes | 5
  21 month: No | 10
  24 month: number analyzed (Participants) | 10
  24 month: Yes | 3
  24 month: No | 7

29. Primary Outcome: Caregiver Change in Option and Practice: School Attendance
Description: Participant will be asked the attendance question in survey. It will be answered in Yes/No.
  * Currently, is child attending school in-person, either full-time or as part of a hybrid or part-time schedule? Y/N
  * This question was only asked to caregivers.
  * Caregivers with multiple children enrolled completed a survey for each child.
Time Frame: Baseline, 3 month, 6 month, 9 month, 15 month, 18 month, 21 month, 24 month
Population: The number analyzed varies per row due to varied response rates per question at each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Parent/Child With Children With Medical Complexity (CMC)
Number analyzed (Participants) | 47
Participants
  Baseline: number analyzed (Participants) | 40
  Baseline: Yes | 38
  Baseline: No | 2
  3 month: number analyzed (Participants) | 30
  3 month: Yes | 29
  3 month: No | 1
  6 month: number analyzed (Participants) | 27
  6 month: Yes | 25
  6 month: No | 2
  9 month: number analyzed (Participants) | 18
  9 month: Yes | 17
  9 month: No | 1
  15 month: number analyzed (Participants) | 8
  15 month: Yes | 8
  15 month: No | 0
  18 month: number analyzed (Participants) | 8
  18 month: Yes | 8
  18 month: No | 0
  21 month: number analyzed (Participants) | 17
  21 month: Yes | 17
  21 month: No | 0
  24 month: number analyzed (Participants) | 10
  24 month: Yes | 10
  24 month: No | 0

30. Primary Outcome: Caregiver Change in Option and Practice: Option to Attend School
Description: Participant will be asked the attendance question in survey. It will be answered in Yes/No
  * Currently, if participant wanted, could the child attend school in-person, either full-time or as part of a hybrid or part-time schedule?
  * Survey branching logic asked this question only to participants whose child was not currently attending school in person, either full-time or as part of a hybrid or part-time schedule. The number analyzed represents the number of participants that answered this question.
  * This question was only asked to caregivers.
  * Caregivers with multiple children enrolled completed a survey for each child.
Time Frame: Baseline, 3 month, 6 month, 9 month, 15 month, 18 month, 21 month, 24 month
Population: The number analyzed varies per row due to varied response rates per question at each time point.
  This question is only asked to participants who indicate that their child is not currently attending school. In this aim, few to no participants were asked this question.
  Only 2 participants were asked this question in Aim 1b.
Measure: Count of Participants; unit: Participants
Arm/Group | Parent/Child With Children With Medical Complexity (CMC)
Number analyzed (Participants) | 2
Participants
  Baseline: number analyzed (Participants) | 1
  Baseline: Yes | 1
  Baseline: No | 0
  3 month: number analyzed (Participants) | 1
  3 month: Yes | 1
  3 month: No | 0
  6 month: number analyzed (Participants) | 1
  6 month: Yes | 1
  6 month: No | 0
  9 month: number analyzed (Participants) | 1
  9 month: Yes | 1
  9 month: No | 0
  15 month: number analyzed (Participants) | 0
  15 month: Yes | 0
  15 month: No | 0
  18 month: number analyzed (Participants) | 0
  18 month: Yes | 0
  18 month: No | 0
  21 month: number analyzed (Participants) | 0
  21 month: Yes | 0
  21 month: No | 0
  24 month: number analyzed (Participants) | 0
  24 month: Yes | 0
  24 month: No | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected during active study participation (from 5/2021 to 6/2023); any reportable events are followed to completion. Participants were assessed from enrollment to study exit, an average of two years. Caregivers were not followed for adverse events.
Description: Per protocol, information indicating an undesirable experience with study participation was reported to PI to determine if it's associated with the study. Associated events were reported to the IRB per local guidelines: https://irb.wisc.edu/wp-content/uploads/sites/2/sites/2/2022/07/AEdecisionguidewithFDAVAupdate_10_31_17.pdf. Additionally, events are documented in study files as Note-to-File. All SAEs and study-associated AEs are reported. Non-study related AEs were not collected or reported.
Arm/Group | Children With Medical Complexity (CMC) | School Staff
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/24
Other Adverse Events (participants affected / at risk) | 0/47 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-01-26): https://cdn.clinicaltrials.gov/large-docs/45/NCT04899245/Prot_SAP_001.pdf
  • Informed Consent Form (2022-11-21): https://cdn.clinicaltrials.gov/large-docs/45/NCT04899245/ICF_000.pdf